CLINICAL TRIAL: NCT06756230
Title: Effects of Downhill Walking in Pulmonary Rehabilitation for Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Downhill Walking in IPF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eccentric_IPF
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: IPF; eccentric exercise training; pulmonary rehabilitation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Downhill Walking PR Group (Active Comparator): A standard pulmonary rehabilitation (PR) exercise program will be implemented. Downhill treadmill walking will be included during walking sessions.
  Interventions: Other: Pulmonary Rehabilitation; Other: Downhill Walking
- Standard PR group (Active Comparator): A standard pulmonary rehabilitation (PR) exercise program will be implemented. Walking will be performed on a treadmill without incline.
  Interventions: Other: Pulmonary Rehabilitation; Other: Treadmill Walking without incline

INTERVENTIONS:
Other: Pulmonary Rehabilitation — 8 weeks, 2 sessions per week,
  Aerobic training will be provided as treadmill walking. It will be performed either downhill or on a flat treadmill, depending on the group.
  Warm-up and stretching exercises
  Resistance exercises will be performed with a load equivalent to 50% of 1 maximum repetition. 10 repetitions will be performed in sets, one set in each session. Based on the differences in the general condition of the patients, different workloads and modifications will be used when creating an exercise program for each patient. Resistance exercises will focus on both upper and lower extremity muscles.
Other: Downhill Walking — Treadmill exercise will be applied for 30 minutes in the target heart rate range of 60-80% intensity. The target heart rate method will be used to determine the exercise intensity. Blood pressure, heart rate and Borg Perceived Exertion Scale scores will be monitored during the exercises. Downhill walking training will continue with a constant -10% incline.
  Arms: Downhill Walking PR Group
Other: Treadmill Walking without incline — Treadmill exercise will be applied for 30 minutes in the target heart rate range of 60-80% intensity. The target heart rate method will be used to determine the exercise intensity. Blood pressure, heart rate and Borg Perceived Exertion Scale scores will be monitored during the exercises. Traditional walking training will initially involve walking with a neutral incline.
  Arms: Standard PR group

SUMMARY:
In this study; will examine the effects of downhill walking (eccentric exercise training) on exercise capacity, quality of life, and blood lactate levels in individuals with IPF. After the initial assessment, patients will be randomized into two groups: downhill walking PR group and Standard PR Group.

DETAILED DESCRIPTION:
Individuals diagnosed with idiopathic pulmonary fibrosis who come to the Pulmonary Rehabilitation Unit of Istanbul Süreyyapaşa Chest Diseases and Chest Surgery Education and Research Hospital will be included in this study. Those who meet the inclusion criteria will be randomized into two groups: Downhill Walking Pr Group (n=17) and Standard Pr Group (n=17). Patients will have exercise sessions twice a week for 8 weeks. Patients will be evaluated immediately before the rehabilitation program and the end of 8 weeks exercise programme. In our study, downhill walking training will differ from traditional walking training only in terms of treadmill training protocol. Traditional walking training involves walking on a motorized treadmill with a neutral incline, progressing with increases in speed, while downhill walking training will be performed at a constant -10% incline.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of IPF according to the clinical diagnostic criteria of the American Thoracic Society and/or the European Respiratory Society (ATS-ERS).
* Being between the ages of 18 and 75.
* Being able to walk on a treadmill.
* Having the ability to cooperate.
* No change in current medication in the last month.
* Not participating in a structured activity program for at least six months.
* Accepting the purpose and method of this study voluntarily and give informed consent for the study.

Exclusion Criteria:

* Presence of physical or mental impairment that prevents informed consent or compliance with the protocol.
* Inability to attend more than 20% of pulmonary rehabilitation sessions.
* Presence of major cardiovascular disease (coronary artery disease, uncontrolled hypertension, arrhythmias, or heart failure).
* Presence of existing orthopedic and neuromuscular exercise limitations.
* Acute exacerbation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
6 Minutes Walking Distance (6MWD) | Baseline and the end of the 8 weeks exercise program
  6 MWD means the distance the patient walked in 6 minute walk test. Its unit is meters.
Saint George Quality of life questionnaire | Baseline and the end of the 8 weeks exercise program
  The St. George's Respiratory Questionnaire (SGRQ) is designed to measure quality of life. Four scores are calculated Symptoms, Activity, Impacts, and Total. Saint George Respiratory Questionaire (SGRQ) score: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).

SECONDARY OUTCOMES:
Spirometric measurements (Forced vital capacity) | Baseline and the end of the 8 weeks exercise program
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. Forced vital capacity (FVC): the maximum amount of air that can be forcibly exhaled from the lungs after fully inhaling. It can be recorded in percentages or liters.
Spirometric measurements (First second forced expiratory volume) | Baseline and the end of the 8 weeks exercise program
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. First-second forced expiratory volume (FEV1): the amount of air that can be exhaled with force in 1 second. It can be recorded in percentages or liters.
Spirometric measurements (FEV1/FVC ratio) | Baseline and the end of the 8 weeks exercise program
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. It is calculated by dividing FEV1 by FVC. It is expressed as a percentage.
Peripheral muscle strength | Baseline and the end of the 8 weeks exercise program
  Peripheral muscle strength will be assessed using a digital dynamometer. Quadriceps femoris muscle strength; will be measured by applying maximum resistance 2-3 cm above the ankle malleolus of the patients in a sitting position using an digital dynamometer.
Hand grip strength | Baseline and the end of the 8 weeks exercise program
  Hand grip strength will be assessed in a sitting position. During the test, the arm will be measured next to the body, with the shoulder adducted, the elbows flexed at 90°, the forearm and wrist in a neutral position, and patients will be asked to grip and release the dynamometer as strongly as possible, and the measurement will be repeated 3 times on both dominant and non-dominant extremities and the averages will be recorded. A one-minute rest will be given between each trial.
Modified Medical Research Council Dyspnea Score | Baseline and the end of the 8 weeks exercise program
  Modified Medical Council Dyspnea score will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4point" means severe dyspnea perception.
Fatigue severity scale | Baseline and the end of the 8 weeks exercise program
  Fatigue levels of individuals will be assessed with the Fatigue Severity Scale (FSS). The FSS consists of 9 questions scored using a 7-point Likert scale, indicating a perception of fatigue that may require medical intervention.
Hospital anxiety depression scale (HADS) | Baseline and the end of the 8 weeks exercise program
  A scale consisting of 14 items developed by Zigmond and Snaith. Seven of these items evaluate anxiety symptoms and seven evaluate depression symptoms. The items in the scale are evaluated with a 4-point Likert scale and are based on a scoring system between 0-3.
Determination of blood lactate level | Baseline and the end of the 8 weeks exercise program
  Blood lactate level will be measured by fingertip sample using a portable lactate meter after a standardized exercise protocol applied before and after the intervention. Blood samples will be recorded in mmol/L after being analyzed by the device.
Carbon monoxide diffusion capacity | Baseline and the end of the 8 weeks exercise program
  Carbon monoxide diffusion capacity (DLCO) is the measurement of the passage of carbon monoxide gas in inspired air into the lung capillary blood. Diffusion test is performed in the pulmonary function test laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No